CLINICAL TRIAL: NCT04875962
Title: A Double-Blind, Placebo-Controlled, Multiple Dose Study to Evaluate Safety, Tolerability, and Pharmacokinetics of UCB0599 in Healthy Study Participants and Patients With Parkinson's Disease (PD)
Brief Title: A Study to Test the Safety, Tolerability, and Pharmacokinetics of UCB0599 in Healthy Study Participants and Patients With Parkinson's Disease (PD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: UCB Biopharma S.P.R.L. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UP0077
Record Dates: First submitted 2021-05-03; First posted 2021-05-06 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Parkinson's Disease
Keywords: UCB0599; Parkinson's Disease; Phase 1 study; Healthy participants; Patients
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1 - UCB0599 (Experimental): Participants will be randomized to receive a predefined dosage of UCB0599.
  Interventions: Drug: UCB0599
- Cohort 2 - UCB0599 (Experimental): Participants will be randomized to receive a predefined dosage of UCB0599.
  Interventions: Drug: UCB0599
- Cohort 1 - Placebo (Placebo Comparator): Participants will be randomized to receive a predefined dosage of Placebo.
  Interventions: Drug: Placebo
- Cohort 2 - Placebo (Placebo Comparator): Participants will be randomized to receive a predefined dosage of Placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: UCB0599 — Participants will receive an assigned dosage regimen of UCB0599 during the Treatment Period.
  Arms: Cohort 1 - UCB0599; Cohort 2 - UCB0599
Drug: Placebo — Participants will receive an assigned dosage regimen of Placebo during the Treatment Period to maintain the blinding.
  Arms: Cohort 1 - Placebo; Cohort 2 - Placebo

SUMMARY:
The purpose of the study is to evaluate the safety and tolerability after administration of multiple doses and the pharmacokinetics (PK) of single and multiple doses of UCB0599 in healthy study participants and participants with Parkinson's Disease (PD).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be 40 to 80 years of age inclusive, at the time of signing the informed consent
* Study participant with Parkinson's disease (PD) must have a clinical diagnosis of PD. The following diagnostic criteria must be met: Bradykinesia AND at least ONE of the following: muscular rigidity or resting tremor
* Study participant with PD must have a historic brain image (magnetic resonance imaging (MRI) or computerized tomography (CT) obtained at any point from the time of clinical diagnosis to the time of Screening that does not show any brain abnormalities that could cause symptomatic Parkinsonism
* Study participant must have a Hoehn and Yahr Stage: 1 to 3
* Study participant must be either untreated, or treated with a stable regimen (at least 4 weeks prior to Baseline Visit) of antiparkinsonian drugs and is expected to remain on this regimen for the duration of the study
* Body weight >50 kg (110 lbs) and body mass index (BMI) within the range 18 to 32 kg/m^2 (inclusive)

Exclusion Criteria:

* Study participant has a known hypersensitivity to any components of the study medication or comparative drugs as stated in this protocol
* Study participant has a known relevant allergy, a pre-existing history of a relevant allergic condition, or a predisposition for an allergic reaction (ie, total immunoglobulin E [IgE] value above normal range at Screening); this study participant's inclusion should be discussed with the Medical Monitor
* Study participant has a history of levodopa-induced motor fluctuations or dyskinesia expected to interfere with his/her ability to participate in the study
* Study participant has ongoing significant inflammatory gastrointestinal disorders and/or clinical signs of significant gastrointestinal problems at Screening
* Study participant has a historic brain scan (MRI scan or CT scan) or an MRI scan performed at Screening indicative of a clinically significant abnormality
* Study participant has a diagnosis of a significant Central nervous system (CNS) disease other than PD or history of epilepsy or seizure disorder other than febrile seizures as a child
* Abnormalities in lumbar spine previously known or determined by a screening lumbar x-ray (if conducted)
* History of clinically significant back pain, back pathology, and/or back injury (for example, degenerative disease, spinal deformity, or spinal surgery) that may predispose participant to complications or technical difficulty with lumbar puncture
* Evidence or history of significant active bleeding or coagulation disorder or use of drugs that affect coagulation or platelet function within 14 days prior to lumbar catheter insertion
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Study participant has a history or present condition of respiratory or cardiovascular disorders at Screening (eg, cardiac insufficiency, coronary heart disease, uncontrolled hypertension, arrhythmia, tachyarrhythmia, or myocardial infarction) which is considered clinically significant by the Investigator
* Study participant has medical history or current diagnosis of diabetes
* Study participant has clinical significant electrocardiogram (ECG) abnormality at Screening, in the opinion of the Investigator
* Study participant has had prior treatment with an investigational vaccine for PD (including active immunization or passive immunotherapy with monoclonal antibodies)
* Study participant has had prior surgical treatment of PD involving intracranial surgery or implantation of a device (including deep brain stimulation) or duodopa

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2019-05-06 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-19 (Actual)

PRIMARY OUTCOMES:
Treatment-Emergent Adverse Avents (TEAEs) from Baseline to End of Study visit | From Baseline to End of study visit (up to Week 7)
  An Adverse Event (AE) is any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product, which does not necessarily have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) in healthy participants on Day 1 | Day 1: Predose up to 12 hours post dose
  Cmax: Maximum observed plasma concentration
Maximum observed plasma concentration (Cmax) in healthy participants on Day 28 | Day 28: Predose up to 24 hours post dose
  Cmax: Maximum observed plasma concentration
Time to maximum observed plasma concentration (tmax) in healthy participants on Day 1 | Day 1: Predose up to 12 hours post dose
  Tmax: Time of observed Cmax
Time to maximum observed plasma concentration (tmax) in healthy participants on Day 28 | Day 28: Predose up to 24 hours post dose
  Tmax: Time of observed Cmax
Area under the concentration - time curve (AUC(0-12h)) from time 0 to 12 hours in healthy participants on Day 1 | Day 1: Predose up to 12 hours post dose
  AUC(0-12h): Area under the curve from time 0 to 12 hours
Area under the concentration-time curve for the dosing interval (AUCtau) in healthy participants on Day 28 | Day 28: Predose up to 24 hours post dose
  AUCtau: Area under the concentration-time curve for the dosing interval at steady state
Maximum observed plasma concentration (Cmax) in patients on Day 1 | Day 1: Predose up to 12 hours post dose
  Cmax: Maximum observed plasma concentration
Maximum observed plasma concentration (Cmax) in patients on Day 28 | Day 28: Predose up to 24 hours post dose
  Cmax: Maximum observed plasma concentration
Time to maximum observed plasma concentration (tmax) in patients on Day 1 | Day 1: Predose up to 12 hours post dose
  Tmax: Time of observed Cmax
Time to maximum observed plasma concentration (tmax) in patients on Day 28 | Day 28: Predose up to 24 hours post dose
  Tmax: Time of observed Cmax
Area under the concentration - time curve (AUC(0-12h)) from time 0 to 12 hours in patients on Day 1 | Day 1: Predose up to 12 hours post dose
  AUC(0-12h): Area under the curve from time 0 to 12 hours
Area under the concentration-time curve for the dosing interval (AUCtau) in patients on Day 28 | Day 28: Predose up to 24 hours post dose
  AUCtau: Area under the concentration-time curve for the dosing interval at steady state

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273 (UCB)
Locations (6):
- United States (6):
  - Up0077 102, Long Beach, California
  - Up0077 103, Bay Harbor Islands, Florida
  - Up0077 105, DeLand, Florida
  - Up0077 107, Atlanta, Georgia
  - Up0077 101, Farmington Hills, Michigan
  - Up0077 104, Raleigh, North Carolina

IPD SHARING:
Plan to Share IPD: No
Due to the small sample size in this trial, IPD cannot be adequately anonymized i.e., there is a reasonable likelihood that individual participants could be re-identified. For this reason, data from this trial cannot be shared.

REFERENCES:
- [Derived] Mercier J, Bani M, Colson AO, Germani M, Lalla M, Plisson C, Huiban M, Searle G, Mathy FX, Nicholl R, Otoul C, Smit JW, van Asch V, Wagneur M, Maguire RP. Evaluation and Application of a PET Tracer in Preclinical and Phase 1 Studies to Determine the Brain Biodistribution of Minzasolmin (UCB0599). Mol Imaging Biol. 2024 Apr;26(2):310-321. doi: 10.1007/s11307-023-01878-7. Epub 2023 Dec 18. PMID 38110790
- [Derived] Smit JW, Basile P, Prato MK, Detalle L, Mathy FX, Schmidt A, Lalla M, Germani M, Domange C, Biere AL, Bani M, Carson S, Genius J. Phase 1/1b Studies of UCB0599, an Oral Inhibitor of alpha-Synuclein Misfolding, Including a Randomized Study in Parkinson's Disease. Mov Disord. 2022 Oct;37(10):2045-2056. doi: 10.1002/mds.29170. Epub 2022 Aug 12. PMID 35959805